CLINICAL TRIAL: NCT03182946
Title: Correction of Platelet Dysfunction Following Traumatic Brain Injury in Geriatric Patients
Brief Title: Correcting Platelet Dysfunction After Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Carolinas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-16-22E
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2021-09

CONDITIONS: Platelet Dysfunction; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from which platelet function and platelet mitochondrial function will be analyzed, as well as serum markers for mitochondrial function
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Platelet mapping Thromboelastography — These diagnostic tests will be acquired in patients with brain injury, to determine prediction of clinical, functional and psychological outcome.
  Other Names: Platelet mitochondrial respiration; Serum presence of microparticles; Serum presence of cardiolipin; Functional independence measure

SUMMARY:
This study evaluates the impact of platelet transfusion on geriatric patients with platelet dysfunction from Traumatic Brain Injury. The authors hypothesize that patients will recover better if their platelet dysfunction is corrected with platelet transfusion.

DETAILED DESCRIPTION:
The geriatric population is subject to traumatic brain injury, often occurring as a result of falls. This patient population is also often receiving anticoagulants and platelet inhibitors increasing their risk of post-injury hemorrhage. Following Traumatic Brain Injury, even without platelet inhibitor medications, platelets become dysfunctional and are no longer able to assist with clot formation. Therefore risk of hemorrhage is increased, both in the brain, and other hemorrhagic sites. Clinical practice at Carolinas Medical Center is to transfuse platelets in patients with platelet dysfunction following brain injury. The current study is investigating the impact of transfusion on correction of platelet dysfunction and patient outcome.

Furthermore, stored platelet dysfunction can be corrected by supplementation with cytochrome c, which supports mitochondrial function. Therefore, the ability of cytochrome c to correct dysfunction in ex vivo platelets from patients with Traumatic Brain Injury will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Traumatic brain injury with Glasgow Coma Scale Score (GCS) <=13

Exclusion Criteria:

Previously know coagulation dysfunction

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be geriatric patients with moderate to severe TBI (GCS <=13).
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in platelet function | Within 5 hours
  Correction of platelet inhibition measured before and after transfusion through platelet mapping thromboelastography

SECONDARY OUTCOMES:
Mortality | 1-3 months
  Mortality will be compared to admission platelet inhibition
Functional Independence Measure | 6-12 months
  Patient function as measured by Functional Independence Measure compared to platelet inhibition

CONTACTS AND LOCATIONS:
Overall Officials: Susan Evans, MD, Principal Investigator — Carolinas Medical Center
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only collaborators will have patient names for data acquisition.

REFERENCES:
- [Background] Sillesen M, Rasmussen LS, Jin G, Jepsen CH, Imam A, Hwabejire JO, Halaweish I, DeMoya M, Velmahos G, Johansson PI, Alam HB. Assessment of coagulopathy, endothelial injury, and inflammation after traumatic brain injury and hemorrhage in a porcine model. J Trauma Acute Care Surg. 2014 Jan;76(1):12-9; discussion 19-20. doi: 10.1097/TA.0b013e3182aaa675. PMID 24368352
- [Background] Jokar TO, Khalil M, Rhee P, Kulvatunyou N, Pandit V, O'Keeffe T, Tang A, Joseph B. Ratio-based Resuscitation in Trauma Patients with Traumatic Brain Injury: Is There a Similar Effect? Am Surg. 2016 Mar;82(3):271-7. PMID 27099065
- [Background] Ortiz I, Velasco A, Le Borgne S, Revah S. Biodegradation of DDT by stimulation of indigenous microbial populations in soil with cosubstrates. Biodegradation. 2013 Apr;24(2):215-25. doi: 10.1007/s10532-012-9578-1. Epub 2012 Jul 31. PMID 22847399
- [Background] Nekludov M, Bellander BM, Blomback M, Wallen HN. Platelet dysfunction in patients with severe traumatic brain injury. J Neurotrauma. 2007 Nov;24(11):1699-706. doi: 10.1089/neu.2007.0322. PMID 18001200
- [Background] Hukkelhoven CW, Steyerberg EW, Rampen AJ, Farace E, Habbema JD, Marshall LF, Murray GD, Maas AI. Patient age and outcome following severe traumatic brain injury: an analysis of 5600 patients. J Neurosurg. 2003 Oct;99(4):666-73. doi: 10.3171/jns.2003.99.4.0666. PMID 14567601
- [Background] Zharikov S, Shiva S. Platelet mitochondrial function: from regulation of thrombosis to biomarker of disease. Biochem Soc Trans. 2013 Feb 1;41(1):118-23. doi: 10.1042/BST20120327. PMID 23356269
- [Background] Reddoch KM, Pidcoke HF, Montgomery RK, Fedyk CG, Aden JK, Ramasubramanian AK, Cap AP. Hemostatic function of apheresis platelets stored at 4 degrees C and 22 degrees C. Shock. 2014 May;41 Suppl 1(0 1):54-61. doi: 10.1097/SHK.0000000000000082. PMID 24169210
- [Background] Stiegler G, Fischer G, Ramanathan G, Bencur P, Weigel G, Mannhalter C. P-selectin mRNA is maintained in platelet concentrates stored at 4 degrees C. Transfusion. 2009 May;49(5):921-7. doi: 10.1111/j.1537-2995.2008.02073.x. Epub 2009 Jan 21. PMID 19175547
- [Background] Nair PM, Pidcoke HF, Cap AP, Ramasubramanian AK. Effect of cold storage on shear-induced platelet aggregation and clot strength. J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 2):S88-93. doi: 10.1097/TA.0000000000000327. PMID 25159368